CLINICAL TRIAL: NCT00419224
Title: Immunogenicity of Influenza Vaccination (Flu Vac) in Patients Receiving Nonmyeloablative Allogeneic Peripheral Blood Stem Cell Transplantation (NM Allo PBSCT) Compared to Healthy Controls
Brief Title: Influenza Vaccination in Bone Marrow Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4675; RPC 6817
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Influenza
Keywords: Peripheral blood stem cell transplantation; Non-myeloabalative; Influenza vaccination; Humoral immune response; Immunogenicity
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: inactivated split-virus influenza vaccine

SUMMARY:
The purpose of this study is to determine whether influenza vaccination protects patients who receive a certain type of bone marrow transplantation.

DETAILED DESCRIPTION:
Patients who receive bone marrow transplantation are at high risk for complications from influenza infection. It is not whether influenza vaccination protects patients who undergo a type of bone marrow transplantation called "nonmyeloablative", or "reduced intensity" bone marrow transplantation. This study compares the response to influenza vaccination in a group of these patients to that in healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they had received RIC allo HSCT 3 months or more prior to enrollment, and were between the age of 18 and 65 years.
* Controls were health care providers at our institution, between the ages of 18 and 65 years, who were in good health, and who are routinely offered influenza vaccination.

Exclusion Criteria:

* Patients were excluded if they failed to engraft, or had relapse of the underlying disease requiring chemotherapy or immunotherapy.
* Patients and controls were also excluded if they had history of egg allergy, acute febrile illness at the time of vaccination, or influenza-like illness within 4 weeks prior to vaccination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2002-10; Study Completion 2003-04

PRIMARY OUTCOMES:
Is the influenza vaccine immunogenic in patients receiving nonmyeloabalative allogeneic PBSCT compared to healthy controls as judged by their humoral antibody response?

CONTACTS AND LOCATIONS:
Overall Officials: Sherif B Mossad, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States